CLINICAL TRIAL: NCT03907527
Title: Phase I/Ib Study Evaluating Safety and Efficacy of PRGN-3005 UltraCAR-T® (Autologous CAR T Cells) in Advanced Stage Platinum Resistant Ovarian Cancer Patients
Brief Title: Modified Immune Cells (Autologous CAR T Cells) in Treating Patients with Advanced, Recurrent Platinum Resistant Ovarian, Fallopian Tube or Primary Peritoneal Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Precigen, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RG1004303
Record Dates: First submitted 2019-04-05; First posted 2019-04-09 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Platinum-Resistant Fallopian Tube Carcinoma; Platinum-Resistant Ovarian Carcinoma; Platinum-Resistant Primary Peritoneal Carcinoma; Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma; Refractory Fallopian Tube Carcinoma; Refractory Ovarian Carcinoma; Refractory Primary Peritoneal Carcinoma; Stage III Fallopian Tube Cancer AJCC V8; Stage III Ovarian Cancer AJCC V8; Stage III Primary Peritoneal Cancer AJCC V8; Stage IIIA Fallopian Tube Cancer AJCC V8; Stage IIIA Ovarian Cancer AJCC V8; Stage IIIA Primary Peritoneal Cancer AJCC V8; Stage IIIA1 Fallopian Tube Cancer AJCC V8; Stage IIIA1 Ovarian Cancer AJCC V8; Stage IIIA2 Fallopian Tube Cancer AJCC V8; Stage IIIA2 Ovarian Cancer AJCC V8; Stage IIIB Fallopian Tube Cancer AJCC V8; Stage IIIB Ovarian Cancer AJCC V8; Stage IIIB Primary Peritoneal Cancer AJCC V8; Stage IIIC Fallopian Tube Cancer AJCC V8; Stage IIIC Ovarian Cancer AJCC V8; Stage IIIC Primary Peritoneal Cancer AJCC V8; Stage IV Fallopian Tube Cancer AJCC V8; Stage IV Ovarian Cancer AJCC V8; Stage IV Primary Peritoneal Cancer AJCC V8; Stage IVA Fallopian Tube Cancer AJCC V8; Stage IVA Ovarian Cancer AJCC V8; Stage IVA Primary Peritoneal Cancer AJCC V8; Stage IVB Fallopian Tube Cancer AJCC V8; Stage IVB Ovarian Cancer AJCC V8; Stage IVB Primary Peritoneal Cancer AJCC V8
Keywords: Platinum resistant; Ovarian Cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (PRGN-3005 UltraCAR-T cells) IP Administration (Experimental): Patients receive autologous PRGN-3005 UltraCAR-T cells via IP administration with or without lymphodepleting chemotherapy.
  Interventions: Biological: PRGN-3005 UltraCAR-T cells
- Treatment (PRGN-3005 UltraCAR-T cells) IV Administration (Experimental): Patients receive autologous PRGN-3005 UltraCAR-T cells via IV administration with or without lymphodepleting chemotherapy.
  Interventions: Biological: PRGN-3005 UltraCAR-T cells

INTERVENTIONS:
Biological: PRGN-3005 UltraCAR-T cells — Given IP
  Arms: Treatment (PRGN-3005 UltraCAR-T cells) IP Administration
Biological: PRGN-3005 UltraCAR-T cells — Given IV
  Arms: Treatment (PRGN-3005 UltraCAR-T cells) IV Administration

SUMMARY:
This is a Phase I/Ib dose escalation, dose expansion, study to evaluate the safety and identify the recommended dose of modified immune cells PRGN-3005 (autologous chimeric antigen receptor (CAR) T cells developed by Precigen, Inc.) in treating patients with ovarian, fallopian tube, or primary peritoneal cancer that has spread to other places in the body, that has come back and is resistant to platinum chemotherapy. Autologous CAR T cells are modified immune cells that have been engineered in the laboratory to specifically target a protein found on tumor cells and kill them.

ELIGIBILITY:
Inclusion Criteria:

* Women with recurrent, advanced, platinum resistant ovarian, fallopian tube, and primary peritoneal cancer that have progressed after receiving standard of care therapies or are not eligible to receive available therapies with known clinical benefit will be eligible for the study. Patients must have measurable disease that can be accurately measured by RECIST 1.1 criteria in at least one dimension as >= 1.0 cm or > 1.5 cm lymph node with computed tomography (CT), ultrasound, or magnetic resonance imaging (MRI) techniques.

  * Platinum resistant is defined as progression of disease within six months of platinum regimen.
  * Patients with BRCA mutations who have completed standard therapies (including PARP inhibitors) are allowed on this study.
* Patients must be capable of understanding and providing a written informed consent.
* Patients must be 14 days from previous cytotoxic chemotherapy at time of cell collection.
* Laboratory values must indicate adequate organ function.
* Patients must be at least 28 days post systemic steroids prior to enrollment except as premedication for contrast allergy and/or other protocol-mandated medication.
* Patients must have Eastern Cooperative Oncology Group (ECOG) performance status score of =< 2.
* Patients must have recovered from major acute infections and/or recent surgical procedures, and in the opinion of the investigator, not have any significant active concurrent medical illnesses precluding protocol treatment.
* Negative pregnancy test for women of childbearing potential. Women of childbearing potential are those who have not been surgically sterilized, are < 60 years old, or have had menses within the past 12 months.
* Women of childbearing potential must be willing to use 2 methods of contraception before, during, and at least 4 months after the PRGN-3005 cell infusion.

Exclusion Criteria:

* Patients with any of the following cardiac conditions:

  * Symptomatic restrictive cardiomyopathy
  * Unstable angina or symptomatic coronary artery disease within 4 months prior to enrollment
  * New York Heart Association functional class III-IV heart failure on active treatment
  * Symptomatic pericardial effusion
  * Congestive heart failure
  * Clinically significant hypotension.
* Patients with CA 125 =< ULN during screening.
* Patients with history of human immunodeficiency virus (HIV), West Nile, Zika, or active hepatitis B or C infections.
* Patients with severe, symptomatic ascites requiring diuretics, regular paracentesis, or other invasive interventions.
* Patients within 28 days of receiving another investigational agent.
* Patients with pulmonary hypertension, pulmonary fibrosis, or restrictive lung disease, patients with baseline oxygen saturation on room air < 92%, forced expiratory volume in 1 second (FEV1) =< 50%, or diffusion capacity of the lung for carbon monoxide (DLco) (corrected) of < 40% will be excluded.
* Women who are pregnant or breast feeding.
* Patients with second malignancy within the last 5 years excluding basal carcinoma of the skin, squamous carcinoma of the skin, or in situ cervical dysplasia that has undergone curative therapy.
* Patients with an active autoimmune disease requiring immunosuppressive therapy or uncontrolled with treatment.
* Patients who are simultaneously enrolled in any other treatment study.
* Clinical or radiological evidence of acute bowel obstruction within 30 days of signing consent.
* Patients with known or treated brain metastases.
* Patients with an active seizure disorder.
* Any female patient <60 years old who does not meet at least one of the following criteria will be considered to have reproductive potential:

  * Post-menopausal for at least 12 consecutive months (i.e., no menses), or
  * Undergone a sterilization procedure (hysterectomy, salpingectomy, or bilateral oophorectomy; tubal ligation is not considered a sterilization procedure). Pregnancy test for females of reproductive potential must be negative within 14 days before leukapheresis.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Estimated)
Dates: Start 2019-04-30 (Actual); Primary Completion 2024-12-15 (Estimated); Study Completion 2028-11-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 12 months after infusion
  Toxicity grading will be evaluated according to the Cancer Therapy Evaluation Program Common Terminology Criteria for Adverse Events version 5.0 and monitoring of adverse events
Maximal tolerated dose of PRGN-3005 | Up to 28 days
  Will be determined by a 3 X 3 dose escalation study for both intraperitoneal infusion and intravenous infusion of the trial.

SECONDARY OUTCOMES:
Evidence of anti-tumor activity | Up to 5 years
  Graded according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
Number of PRGN-3005 T Cells | Up to 12 months post treatment
  Number of PRGN-3005 T Cells present in patients treated with PRGN-3005

CONTACTS AND LOCATIONS:
Overall Officials: Amy R. Lankford, PhD, Study Director — Precigen, Inc
Locations (2):
- United States (2):
  - National Institutes of Health (NIH), Bethesda, Maryland
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No